CLINICAL TRIAL: NCT03787173
Title: Patient-ventilator Synchronisation Study in Non Invasive Ventilation for Intensive Care Unit Patients: Comparison Between Manual and Automated Ventilator Settings.
Brief Title: Patient-ventilator Synchronisation Study for Intensive Care Unit Patients
Acronym: SyncAutoVNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-CHITS-01; 2018-A00658-47 (Other: Id-RCB)
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Acute Respiratory Failure
Keywords: non invasive ventilation; patient ventilator synchrony; acute respiratory failure; closed loop ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual standard ventilator settings (No Intervention): Inspiratory trigger set at 2 l/min, Expiratory trigger set at 25% of peak inspiratory flow
- Manual optimized ventilator settings (Active Comparator): Inspiratory trigger and Expiratory trigger settings optimized by investigator
  Interventions: Device: Optimized
- Automated ventilator settings (Experimental): Inspiratory trigger and Expiratory trigger settings automatized
  Interventions: Device: Automated

INTERVENTIONS:
Device: Optimized — Inspiratory trigger and Expiratory trigger settings optimized by investigator
  Arms: Manual optimized ventilator settings
Device: Automated — Inspiratory trigger and Expiratory trigger settings automatized
  Arms: Automated ventilator settings

SUMMARY:
This cross-over study will compare the asynchrony index between standard manual ventilator settings, optimized manual ventilator settings, and automated ventilator setting in intensive care patients ventilated in non-invasive ventilation with a high asynchrony index. The hypothesis is that both manual optimized ventilator settings and automated ventilator settings are associated with a lower patient-ventilator asynchrony index as compared to manual standard ventilator settings.

A randomized cross-over design method will be used. Patient requiring NIV with an asynchrony index over 35% will be included. An esophageal catheter with a balloon will be inserted to monitor esophageal pressure. Patients will be ventilated during 3 periods of 30 min, with 10 minutes of washout in between. Recordings of airway pressure, airway flow, and esophageal pressure will be analyzed by two investigators blinded of the trigger settings.

The primary outcome will be the asynchrony index. The secondary outcome will be the ineffective inspiratory effort index, autotrigering index, double triggering index, inspiratory trigger delay, cycling delay, total time spent in asynchrony, patient comfort, and blood gas results.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is used in 35% of patient admitted in intensive care unit (ICU) with a failure rate of 10 to 70% depending on the indication and clinician experience. Patient-ventilator asynchrony is a frequent cause of NIV failure. Therefore, optimizing patient-ventilator synchronization is important for its comfort, tolerance, and efficacy. An optimal patient-ventilation is achieved when the mechanical breath provided by the ventilator match the patient inspiratory effort. The ratio between the number of asynchronies divided by the number of patient inspiratory effort define the asynchrony index (AI). AI over 10% is considered as severe and occurs in 30 to 43% of patients ventilated in NIV. Patient ventilator asynchronies occurs because ventilator settings of inspiratory and expiratory triggers remain constant in patient with variable respiratory drive, and unintentionnals leaks that are difficult to control in NIV. Thus using an automatic adjustment of inspiratory and expiratory triggers setting according to patient effort and unintentional leaks may decrease the number of patient-ventilator asynchronies. This cross-over study will compare the asynchrony index between standard manual ventilator settings, optimized manual ventilator settings, and automated ventilator setting in intensive care patients ventilated in non-invasive ventilation with a high asynchrony index. The hypothesis is that both manual optimized ventilator settings and automated ventilator settings are associated with a lower patient-ventilator asynchrony index as compared to manual standard ventilator settings.

A randomized cross-over design method will be used. Patient requiring NIV with an asynchrony index over 30% will be included. An esophageal catheter with a balloon will be inserted to monitor esophageal pressure. Patients will be ventilated during 3 periods of 30 min, with 10 minutes of washout in between. Recordings of airway pressure, airway flow, and esophageal pressure will be analyzed by two investigators blinded of the trigger settings.

The primary outcome will be the asynchrony index. The secondary outcome will be the ineffective inspiratory effort index, autotrigering index, double triggering index, inspiratory trigger delay, cycling delay, total time spent in asynchrony, patient comfort, and blood gas results.

The sample size was calculated from the total asynchrony index (primary outcome). Patients with an asynchrony index over 30% in using manual standard ventilator settings will be included. Considering an asynchrony index of 30 ± 15 % in manual standard ventilator settings with a clinically significant objective to reduce the asynchrony index to 15% in manual optimized ventilator settings and automated ventilator settings, a sample size of 30 patients is required with a risk at 0.05 and a power at 80%. Therefore, 35 patients are planned.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old
* Covered by social insurance
* Consent for study signed by patient or next-of-kin
* NIV session indicated for at least 2 hours
* Asynchrony index ≥ 30% with standard manual settings

Exclusion Criteria:

* Patient requiring continuous NIV
* Contra-indication to esophageal catheter insertion: gastric ulcer, esophageal varices, pharyngeal or laryngeal tumor.
* Patient with withholding decision about intubation
* Moribund patient
* Patient included in another interventional study in the last 30 days
* Patient that does not speak French
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Asynchrony index | Continuous measurement over 30min
  Ratio between the total number of asynchronies divided by the number of patient inspiratory effort

SECONDARY OUTCOMES:
Lineffective inspiratory effort index | Continuous measurement over 30min
  Ratio between the total number of ineffective inspiratory effort divided by the number of patient inspiratory effort
Autotrigering index | Continuous measurement over 30min
  Ratio between the total number of autotriggered breath divided by the number of patient inspiratory effort
Double triggering index | Continuous measurement over 30min
  Ratio between the total number of double triggered breath divided by the number of patient inspiratory effort
Inspiratory trigger delay | Continuous measurement over 30min
  Time between the beginning of patient effort assessed on oesophageal pressure and beginning of mechanical breath.
Cycling delay | Continuous measurement over 30min
  Time between the end of patient effort assessed on oesophageal pressure and the end of mechanical breath.
Total time spent in asynchrony | Continuous measurement over 30min
  Ratio of total time of ineffective inspiratory effort, inspiratory trigger delay, and cycling delay on total time of recording.
Patient comfort | 1 day (Single measurement)
  Visual analog scale of Likert type measuring patient comfort going from 0 (very uncomfortable) to 10 (very comfortable)
Blood PaO2 results | After each period at 30 min, 1 h and 1 h 30 min
  PaO2
Blood PaCO2 results | After each period at 30 min, 1 h and 1 h 30 min
  PaCO2
Blood pH results | After each period at 30 min, 1 h and 1 h 30 min
  pH

CONTACTS AND LOCATIONS:
Overall Officials: Aude Garnero, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demoule A, Chevret S, Carlucci A, Kouatchet A, Jaber S, Meziani F, Schmidt M, Schnell D, Clergue C, Aboab J, Rabbat A, Eon B, Guerin C, Georges H, Zuber B, Dellamonica J, Das V, Cousson J, Perez D, Brochard L, Azoulay E; oVNI Study Group; REVA Network (Research Network in Mechanical Ventilation). Changing use of noninvasive ventilation in critically ill patients: trends over 15 years in francophone countries. Intensive Care Med. 2016 Jan;42(1):82-92. doi: 10.1007/s00134-015-4087-4. Epub 2015 Oct 13. PMID 26464393
- [Background] Demoule A, Girou E, Richard JC, Taille S, Brochard L. Increased use of noninvasive ventilation in French intensive care units. Intensive Care Med. 2006 Nov;32(11):1747-55. doi: 10.1007/s00134-006-0229-z. Epub 2006 Jun 24. PMID 16799775
- [Background] Keenan SP, Sinuff T, Burns KE, Muscedere J, Kutsogiannis J, Mehta S, Cook DJ, Ayas N, Adhikari NK, Hand L, Scales DC, Pagnotta R, Lazosky L, Rocker G, Dial S, Laupland K, Sanders K, Dodek P; Canadian Critical Care Trials Group/Canadian Critical Care Society Noninvasive Ventilation Guidelines Group. Clinical practice guidelines for the use of noninvasive positive-pressure ventilation and noninvasive continuous positive airway pressure in the acute care setting. CMAJ. 2011 Feb 22;183(3):E195-214. doi: 10.1503/cmaj.100071. Epub 2011 Feb 14. No abstract available. PMID 21324867
- [Background] Ferrer M, Valencia M, Nicolas JM, Bernadich O, Badia JR, Torres A. Early noninvasive ventilation averts extubation failure in patients at risk: a randomized trial. Am J Respir Crit Care Med. 2006 Jan 15;173(2):164-70. doi: 10.1164/rccm.200505-718OC. Epub 2005 Oct 13. PMID 16224108
- [Background] El-Solh AA, Aquilina A, Pineda L, Dhanvantri V, Grant B, Bouquin P. Noninvasive ventilation for prevention of post-extubation respiratory failure in obese patients. Eur Respir J. 2006 Sep;28(3):588-95. doi: 10.1183/09031936.06.00150705. Epub 2006 May 31. PMID 16737982